CLINICAL TRIAL: NCT05637957
Title: The Feasibility of Transcranial Direct Current Stimulation as an Adjunct to Outpatient Physiotherapy in Children With Acquired Brain Injury
Brief Title: Feasibility of tDCS as an Adjunct to Outpatient Physiotherapy in Children With ABI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 504
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Acquired Brain Injury; Stroke; Traumatic Brain Injury; Hemiparesis
Keywords: transcranial direct current stimulation; physiotherapy; pediatric; motor learning
MeSH Terms: conditions — Brain Injuries; Stroke; Brain Injuries, Traumatic; Paresis

STUDY DESIGN:
Intervention Model Description: Parallel group randomized feasibility trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Physiotherapists providing treatment, physiotherapists conducting assessment, research coordinator, principal investigators, participants are all blinded to treatment allocation. Research assistants administered the transcranial direct current stimulation are not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy + Active tDCS (Experimental): 20 minutes of active anodal tDCS immediately prior to physiotherapy intervention, twice a week for total of 10 sessions.
  Interventions: Device: active transcranial direct current stimulation
- Physiotherapy + Sham tDCS (Active Comparator): 20 minutes of sham anodal tDCS immediately prior to physiotherapy intervention, twice a week for total of 10 sessions.
  Interventions: Device: sham transcranial direct current stimulation

INTERVENTIONS:
Device: active transcranial direct current stimulation — Device: 20 minutes of up to 2.0 mA active anodal tDCS (anode positioned at C3/4, cathode positioned at Fp1/2 as per 10-20 electrode placement guidelines) Behavioral: Physiotherapy motor skills based physiotherapy intervention (representative of typical goal-focused intervention in the clinical ABI program at Holland Bloorview), 45 minutes in duration
  Arms: Physiotherapy + Active tDCS
Device: sham transcranial direct current stimulation — Device: 1 minute of 1.0 mA anodal tDCS (anode positioned at C3/4, cathode positioned at Fp1/2 as per 10-20 electrode placement guidelines) and 19 minutes with unit turned off and electrodes remaining in place Behavioral: Physiotherapy motor skills based physiotherapy intervention (representative of typical goal-focused intervention in the clinical ABI program at Holland Bloorview), 45 minutes in duration
  Arms: Physiotherapy + Sham tDCS

SUMMARY:
This study will evaluate the feasibility of transcranial direct current stimulation (tDCS) as an adjunct to an outpatient motor skills-based physiotherapy intervention for children and youth with acquired brain injury. Up to 10 children (age 5-18 years) with childhood onset stroke or traumatic brain injury will be randomly allocated to receive active or sham anodal tDCS immediately prior to the physiotherapy session. These sessions will occur twice weekly for a total of 10 sessions. Assessment of gross motor outcome measures will occur immediately before and after the combined tDCS and physiotherapy treatment protocol. The preliminary treatment effect between the two treatment groups will be compared and other feasibility indicators will be evaluated.

DETAILED DESCRIPTION:
Objectives: The purpose of this study is to evaluate the feasibility of tDCS as a pre-treatment adjunct to outpatient physiotherapy (our outpatient 'physio+tDCS' protocol) for children with stroke or TBI. The primary objective is to evaluate the feasibility of an outpatient twice weekly 'physio+tDCS' protocol given over five weeks, as measured by participant eligibility, recruitment, tolerance, retention, and adherence to treatment protocol (e.g., session frequency and completion timelines). The secondary objective is to explore the preliminary effect of physio+tDCS on gross motor function in children with childhood onset stroke and TBI, as measured by individualized goal achievement and standardized gross motor outcome measures.

Randomization and Blinding: Once enrolled in the study, an independent research assistant (RA) will randomly assign each child to the "sham" or "active" tDCS treatment group using a computer randomization web-based program. Only the RAs involved in the study will be aware of each participant's treatment group assignment. The participants and the assessing/treating PTs will be blinded to the participant's treatment group.

Intervention:

tDCS Treatment- Depending on treatment group allocation, participants will receive 20 minutes of active tDCS or sham tDCS (provided by a trained RA) immediately prior to two physiotherapy sessions each week for a total of 10 sessions. Children and PTs will be blinded to their tDCS/sham allocation. Two electrodes (5x7cm) in size will be used such that the anodal electrode will be attached to the C3/4 position on the scalp, to target the lower extremity region of the primary motor cortex most affected by their brain injury, and the cathodal electrode will be attached to the contralateral supraorbital (Fp1/Fp2) area of the forehead. Each tDCS treatment will consist of up to 2.0 mA of stimulation, adjusting for the child's age, head size, and tolerance as required. Participant symptoms and safety will be tracked before, during, and after each tDCS session. Adverse events reported via a REB-approved standard process to an independent in-house safety monitoring committee. Physiotherapy Intervention- The physiotherapy treatment paired with the tDCS consists of the typical motor skills-based physiotherapy children receive brain injury program at Holland Bloorview. Each 45-minute physiotherapy session promotes motor learning by focusing on functional tasks related to the child's personalized motor goals. Therapists individualize the program by adapting the tasks, instructions, feedback, and the level of challenge based on the child's needs.

Outcomes Feasibility- Feasibility of study implementation and tDCS will be evaluated by tracking process, resource, and treatment indicators. A priori feasibility targets are as follows: 30% of children indentified by the child's clinical physiotherapist or nurse will be eligible for the study, 70% of eligible children will be recruited; 80% of the tDCS sessions started will last the entire 20-minute duration, 75% of treatment sessions will be completed, and 90% of reassessments will occur in the 14 days following the final treatment session. Adherence to the study protocol will be tracked by the number of tDCS and physiotherapy sessions scheduled per week and the number actually completed. Reasons for cancelled sessions or decreased number of sessions booked will be documented. Because tDCS should optimally occur in the half hour prior to physiotherapy, the start time and duration of stimulation will be documented, as well as the start time and duration of each physiotherapy session, on tracking sheets that will be completed by the RA/therapist conducting each tDCS/physiotherapy session.

Gross Motor- Baseline assessments will be conducted by a blinded independent PT assessor in the two weeks prior to beginning the study treatment protocol. The reassessment will be conducted by the same blinded PT assessor up to two weeks after their last study intervention session. A priori targets for the co-primary gross motor outcomes are as follows: The active tDCS group should have at least 3 mean points of change more than the sham group on the Gross Motor Function Measure (GMFM) and at least 2.0 mean points of change more than the sham group on the Canadian Occupational Performance Measure (COPM).

ELIGIBILITY:
Inclusion Criteria:

* Stroke or moderate to severe traumatic brain injury, diagnosed with imaging (e.g., MRI, CT scan);
* 5-18 years of age inclusive (at time of study enrolment);
* In the outpatient stage of rehabilitiation
* Followed by a physician through ABI medical follow-up clinic at Holland Bloorview OR previously admitted to the inpatient ABI program at Holland Bloorview;
* Medically stable, as determined by their ABI physician;
* Walks a minimum of 10m with or without assistance;
* Stands independently for 10s;
* Balances for less than 20s on most affected leg;
* Hemiplegia, identified by decreased selective motor control at one ankle compared to the other (i.e., decreased ability to isolate ankle plantar flexion and dorsiflexion on the more affected ankle);
* Available to attend twice weekly appointments for five weeks, as well as a two-hour baseline and post-treatment assessment;
* Tolerates 2 hours of physiotherapy assessment (with short breaks as needed);
* Tolerates 45 minutes of physiotherapy treatment;
* Capable of participating in standardized physiotherapy assessment, from a cognitive and behavioural perspective; and
* Can communicate discomfort either verbally or non-verbally
* Follows directions provided in English
* Parent/legal guardian can read and speak English

Exclusion Criteria:

* Admitted to acute care or inpatient rehabilitation hospital
* Seizure(s) in the last 6 months;
* Planned medication changes during study (i.e., any medication that affects their ability to participate in therapy from a physical, cognitive, emotional standpoint);
* Botox injections in the last 3 months;
* Brain tumour;
* Metal implants or fragments in the head;
* Cranial bone flap removed;
* Stitches/staples on the head;
* Wounds or unhealed incisions at electrode placement sites;
* Cochlear implant;
* Implanted neurostimulator (e.g., vagal nerve stimulator, deep brain stimulator);
* Cardiac pacemaker;
* Battery-powered medication infusion device (e.g., baclofen or insulin pump);
* Pregnancy;
* Diagnosed with another neuromotor disorder(s) affecting gross motor function (e.g., cerebral palsy, spinal cord injury, etc.…);
* Onset of ABI before the age of two years;
* Neurodegenerative diagnosis;
* Lower extremity weight bearing activity restrictions secondary to injuries (e.g., fracture, ligamentous injury) as present at time of study enrollment;
* Non-orthopaedic activity restrictions that limit gross motor activity (e.g., splenic laceration with orders not to run or jump); or
* Enrolment in another treatment-based research study during the current study

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM-88) | Change from baseline to reassessment (4-6 weeks)
  A standardized physiotherapy assessment (validated for children with ABI) that assesses gross motor function in five dimensions (A- lying & rolling, B- sitting, C- crawling & kneeling, D- standing, walking, E-running & jumping). Each of the 88 items is scored from 0-3.
Canadian Occupational Performance Measure (COPM) | Change from baseline to reassessment (4-6 weeks)
  The Canadian Occupational Performance Measure is a standardized outcome measure that allows children and families to set goals and evaluate their performance and satisfaction with each goal on a scale of 1 to 10, where higher ratings mean increased performance and satisfaction. In this study, the goals will be participation-based goals related to gross motor activities.
Eligibility Rate | Duration of study (approximately 2 years)
  The proportion of eligible participants compared to the number of children identified by brain injury clinicians using preliminary screening checklist.
Enrollment Rate | Duration of study (approximately 2 years)
  The proportion of eligible participants who enrollment in the study.
Adherence Rate | Duration of study (approximately 2 years)
  Proportion of participants who completed 10 treatment sessions
Transcranial direct current stimulation tolerance | Duration of study (approximately 2 years)
  The proportion of tDCS sessions that were started lasting the entire treatment session

SECONDARY OUTCOMES:
Acquired Brain Injury Challenge Assessment (ABI-CA) | Change from baseline to reassessment (4-6 weeks)
  An 18-item standardized assessment of high level gross motor skills in children and youth with ABI. Each item assesses the child's ability to perform a skill and is scored on a 5-point scale according to time and quality of movement (where '5' indicates normal quality of movement and/or completion within a minimum amount of time while '0' indicates they were unable to complete the item within a maximum period of time and did not meet the criteria for quality).
10m Fast Walk Test | Change from baseline to reassessment (4-6 weeks)
  Timed walk test over 10m with the participant walking as fast as possible.
Goal Attainment Scaling | Change from baseline to reassessment (4-6 weeks)
  Participant-specific mobility, balance, and/or gross motor goals created by the treating physiotherapist to target specific activities they will work on in physiotherapy. The child's baseline ability is scored as a '-2'. The physiotherapist sets individualized targets for the child where '-1' indicates they are performing somewhat less than expected, '0' indicates they are performing at the expected level for a given time frame, '+1' indicates they have done somewhat better than expected, and '+2' indicates they have done much better than expected. When the goal is set, the physiotherapist sets '0' (the expected level) based on the timing of the reassessment and what they think the child is clinically capable of accomplishing in that time period.
Pediatric Evaluation of Disability Inventory (Mobility and Self-Care domains) | Change from baseline to reassessment (4-6 weeks)
  Parent-reported computerized questionnaire evaluating their child's function ability. Each item is rated on 4-point scale where '0' indicates the child is unable to do and '4' indicates the activity is easy to do. A higher score indicates higher levels of independence with mobility and self-care.

CONTACTS AND LOCATIONS:
Overall Officials: Deryk Beal, PhD, Principal Investigator — Clinician Scientist; Virginia Wright, PhD, Principal Investigator — Clinician Scientist
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
At this time data will not be shared with other researchers